CLINICAL TRIAL: NCT05230576
Title: Deep Learning Model Based on Routine Ultrasound Scanning Video to Help Doctors Improve the Diagnosis of Carotid Plaque
Brief Title: Intelligent Detection of Carotid Plaque and Its Stability Based on Deep Learning Dynamic Ultrasound Scanning
Status: Completed | Type: Observational
Sponsor: Jia Liu (Other)
Responsible Party: Sponsor-Investigator, Jia Liu, Attending Physician, Department of Ultrasound, The Third Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: [2020]02-255-01
Record Dates: First submitted 2022-01-27; First posted 2022-02-09 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deep learning training cohort: 2/3 of the enrolled patients and their corresponding carotid artery dynamic scan images and expert diagnosis results were randomly selected as the training cohort for deep learning.
  Interventions: Diagnostic Test: Deep learning training cohort
- Deep learning validation cohort: The carotid artery dynamic scan images and expert diagnosis results of the remaining 1/3 patients were used as a validation cohort to evaluate the overall diagnostic accuracy of the deep learning model.
  Interventions: Diagnostic Test: Deep learning validation cohort

INTERVENTIONS:
Diagnostic Test: Deep learning training cohort — train the deep learning model
  Groups: Deep learning training cohort
Diagnostic Test: Deep learning validation cohort — evaluate the model
  Groups: Deep learning validation cohort

SUMMARY:
This study intends to build a model through deep learning that can automatically and accurately detect plaques, calculate the lumen stenosis rate and evaluate the stability of plaques based on the carotid transverse axis dynamic ultrasound images and contrast-enhanced ultrasound images, so as to comprehensively evaluate the possibility of carotid plaques. cardiovascular risk. The successful development of this study will automatically simulate and reproduce the whole process of carotid plaque assessment by clinical sonographers. Solve the problem of ultrasonic inspection equipment and experience dependence. It is expected to carry out large-scale population intelligent screening, providing new ideas for early prevention and treatment. Especially in medically underdeveloped remote areas and the lack of experienced sonographers, it has great practical value in clinical health care and can bring greater social and economic benefits.

DETAILED DESCRIPTION:
Background:

Carotid plaque is harmful to human health. According to estimates by the World Health Organization, 6.7 million cerebrovascular accidents and strokes occur each year, mainly related to the formation of carotid atherosclerotic plaques. On the one hand, carotid artery plaque can cause carotid artery stenosis or even occlusion, causing cerebral ischemia. Early detection and accurate assessment of carotid plaques are helpful for clinicians to take effective intervention measures, which can significantly reduce the disability rate and fatality rate of stroke.

Carotid CTA and MRA can provide relatively high-resolution and high-quality plaque images, but have cost and scanning limitations that limit their application in daily clinical practice. Ultrasonography has the advantages of non-invasiveness, convenience, low cost, and good repeatability. It is the preferred imaging method for plaque detection, stenosis and plaque stability. Contrast-enhanced ultrasonography (CEUS) can sensitively demonstrate intra-plaque microcirculation perfusion by injecting microbubble contrast agents, and is consistent with histopathological findings, and has been increasingly used clinically to evaluate plaque stability.

However, on the one hand, the limitation of ultrasound examination is that it needs to rely on the level of instruments and operators to improve the accuracy. On the other hand, with the growth of the population base and the aging of society, the traditional medical model has been unable to meet the annual increase in the number of patients. examination needs of patients. Therefore, it is of great significance to develop an integrated AI application platform that can automatically and accurately detect plaque based on ultrasound image data, and evaluate lumen stenosis and plaque stability.

Purpose:

This study intends to build a model based on deep learning to automatically and accurately detect plaque based on the carotid transverse axis dynamic ultrasound image, calculate the lumen stenosis rate, and perform stability assessment, so as to comprehensively evaluate the possible cardiovascular effects of carotid plaque. risk. It will realize the automatic simulation and reproduction of the whole process of assessment of cervical plaque by clinical ultrasound experts.

Study design:

Two-thirds of the enrolled patients and their corresponding carotid artery dynamic scan images and expert diagnosis results were randomly selected as the deep learning training cohort. The carotid artery dynamic scan images and expert diagnosis results of the remaining 1/3 patients were used as a validation cohort to evaluate the overall diagnostic accuracy of the deep learning model

Statistical Analysis:

The sensitivity, specificity, positive predictive value, and negative predictive value of deep learning for detecting plaque, estimating luminal stenosis rate, or predicting plaque stability were calculated by the area under the receiver operating characteristic (ROC) curve (AUROC) to evaluate. Statistical analysis was performed using SPSS 22.0 software.

Quality Control:

Develop standardized and standard carotid ultrasound examination methods and operating procedures, and develop unified image acquisition and storage standards. All operators are rigorously trained in carotid ultrasonography. Two operators with more than 5 years of experience in ultrasound operation were hired as quality control personnel to review all images and exclude unqualified images.

Ultrasound is safe and radiation-free. During the examination, the doctor and the patient were always in a state of communication, and the patient felt less nervous and fearful, with good tolerance and high compliance.

Ethics of the study:

This research will follow the ethical guidelines of the Declaration of Helsinki of the World Medical Congress and the relevant norms and regulations of clinical research. The study will begin after the approval of the ethics committee. Before the start of the study, the investigator should inform the subjects of all relevant contents of the clinical study in easy-to-understand language, and inform the patients that they have the right to withdraw from the study at any time. The study was started only after the patients signed the informed consent voluntarily.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age≥18 years old, gender is not limited. (2) Patients who voluntarily participated in this study signed the informed consent.

Exclusion Criteria:

* (1) Severe cerebrovascular disease, uncooperative patients, and those who cannot tolerate examination. (2) Wound dressings after neck surgery affects carotid artery ultrasonography. (3) The neck is short and thick, and the probe cannot be put down vertically.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age≥18 years old, gender is not limited, with varying degrees of carotid atherosclerosis.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
AI assists junior radiologists to read images, and primary physicians read images independently | through study completion, an average of 2 years
  Taking the reading results of senior sonographers as the gold standard, the sensitivity, specificity, accuracy, positive predictive value, and negative predictive value of AI-assisted reading and independent reading by junior physicians for carotid plaque-assisted diagnosis were tested. AUC is evaluated.
Assessing the performance of AI model | through study completion, an average of 2 years
  Taking the reading results of senior sonographers as the gold standard, the sensitivity, specificity, accuracy, positive predictive value, and negative predictive value of AI independent reading. It was evaluated by the area under the receiver operating characteristic (ROC) curve (AUC).
AI estimates the lumen stenosis rate | through study completion, an average of 2 years
  Taking the reading results of senior sonographers as the gold standard, AI can estimate the sensitivity, specificity, accuracy, positive predictive value and negative predictive value of lumen stenosis rate. It was evaluated by the area under the receiver operating characteristic (ROC) curve (AUC).
AI predicts plaque stability. | through study completion, an average of 2 years
  Taking the reading results of senior sonographers as the gold standard, AI predicts the sensitivity, specificity, accuracy, positive predictive value and negative predictive value of plaque stability. It was evaluated by the area under the receiver operating characteristic (ROC) curve (AUC).
Plaque detection by AI model on videos acquired by different types of equipment. | through study completion, an average of 2 years
  Taking the reading results of senior sonographers as the gold standard, AI detects plaque sensitivity, specificity, accuracy, positive predictive value, and negative predictive value on different ultrasound equipment. Assessed by the area under the receiver operating characteristic (ROC) curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Jia Liu, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbott AL, Paraskevas KI, Kakkos SK, Golledge J, Eckstein HH, Diaz-Sandoval LJ, Cao L, Fu Q, Wijeratne T, Leung TW, Montero-Baker M, Lee BC, Pircher S, Bosch M, Dennekamp M, Ringleb P. Systematic Review of Guidelines for the Management of Asymptomatic and Symptomatic Carotid Stenosis. Stroke. 2015 Nov;46(11):3288-301. doi: 10.1161/STROKEAHA.115.003390. Epub 2015 Oct 8. PMID 26451020
- [Background] Nighoghossian N, Derex L, Douek P. The vulnerable carotid artery plaque: current imaging methods and new perspectives. Stroke. 2005 Dec;36(12):2764-72. doi: 10.1161/01.STR.0000190895.51934.43. Epub 2005 Nov 10. PMID 16282537
- [Background] Saba L, Saam T, Jager HR, Yuan C, Hatsukami TS, Saloner D, Wasserman BA, Bonati LH, Wintermark M. Imaging biomarkers of vulnerable carotid plaques for stroke risk prediction and their potential clinical implications. Lancet Neurol. 2019 Jun;18(6):559-572. doi: 10.1016/S1474-4422(19)30035-3. Epub 2019 Apr 4. PMID 30954372
- [Background] Rafailidis V, Charitanti A, Tegos T, Destanis E, Chryssogonidis I. Contrast-enhanced ultrasound of the carotid system: a review of the current literature. J Ultrasound. 2017 Feb 9;20(2):97-109. doi: 10.1007/s40477-017-0239-4. eCollection 2017 Jun. PMID 28592999
- [Background] Deyama J, Nakamura T, Takishima I, Fujioka D, Kawabata K, Obata JE, Watanabe K, Watanabe Y, Saito Y, Mishina H, Kugiyama K. Contrast-enhanced ultrasound imaging of carotid plaque neovascularization is useful for identifying high-risk patients with coronary artery disease. Circ J. 2013;77(6):1499-507. doi: 10.1253/circj.cj-12-1529. Epub 2013 Mar 22. PMID 23519900
- [Background] Varetto G, Gibello L, Castagno C, Quaglino S, Ripepi M, Benintende E, Gattuso A, Garneri P, Zan S, Capaldi G, Bertoldo U, Rispoli P. Use of Contrast-Enhanced Ultrasound in Carotid Atherosclerotic Disease: Limits and Perspectives. Biomed Res Int. 2015;2015:293163. doi: 10.1155/2015/293163. Epub 2015 Jun 21. PMID 26180793
- [Background] Staub D, Patel MB, Tibrewala A, Ludden D, Johnson M, Espinosa P, Coll B, Jaeger KA, Feinstein SB. Vasa vasorum and plaque neovascularization on contrast-enhanced carotid ultrasound imaging correlates with cardiovascular disease and past cardiovascular events. Stroke. 2010 Jan;41(1):41-7. doi: 10.1161/STROKEAHA.109.560342. Epub 2009 Nov 12. PMID 19910551